CLINICAL TRIAL: NCT02143050
Title: A Phase I/II Trial of Dabrafenib, Trametinib and Metformin Administered to Unresectable Stage IIIC and Stage IV BRAF V600E + Melanoma Patients
Brief Title: Study of Dabrafenib, Trametinib and Metformin for Melanoma Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No participant enrollment
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Jason Chesney, Director, James Graham Brown Cancer Center, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCC-MEL-14-01
Record Dates: First submitted 2014-05-13; First posted 2014-05-20 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Melanoma
Keywords: Unresectable melanoma Stage IIIC and Stage IV BRAF V600E+
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dabrafenib, Trametinib and Metformin (Experimental): Dabrafenib 150 mg PO BID until progression or unacceptable toxicity. Trametinib 2 mg PO QD until progression or unacceptable toxicity. Metformin 500 mg PO BID x 2 weeks, then 850 mg PO BID until progression or unacceptable toxicity.
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Drug: Metformin

INTERVENTIONS:
Drug: Dabrafenib
  Other Names: Tafinlar
Drug: Trametinib
  Other Names: Mekinist
Drug: Metformin
  Other Names: Glucophage

SUMMARY:
The main purpose is to evaluate the clinical response, safety and survival of the FDA approved drugs Dabrafenib, Trametinib in combination with Metformin. Investigators hypothesize that the combination of an FDA approved non toxic dose of oral Metformin with the B-Raf inhibitor, Dabrafenib and the MEK inhibitor, Trametinib will yield little toxicity and improve clinical outcomes in terms of objective response rates and survival in metastatic melanoma patients.

DETAILED DESCRIPTION:
The study will be a single-arm, single center, uncontrolled phase I/II trial to estimate the safety of the combined treatments and then estimate the efficacy in terms of objective response rate in patients with stage IIIC and Stage IV melanoma treated with dabrafenib/trametinib and metformin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years of age
* Patients with histologically confirmed BRAFV600E melanoma (Stage IIIC or
* Stage IV, American Joint Commission on Cancer)
* Eastern Cooperative Oncology Group Performance Status of 0 to 2
* Life expectancy > 3 months
* At least 1 site of radiographically measurable disease by RECIST 1.1
* Adequate hematologic, renal, and liver function as defined by laboratory values performed within 42 days prior to initiation of dosing:
* Absolute neutrophil count > 1.0 x 10⁹/L
* Platelet count > 50 x 10⁹/L
* Hemoglobin > 8 g/dL
* Serum creatinine < 2 x upper limit of normal
* Total serum bilirubin < 3 x ULN
* Serum aspartate transaminase or serum alanine transaminase < 3 x ULN, and < 4 x ULN if liver metastases are present
* Fertile males should use an effective method of contraception during treatment and for at least 3 months after completion of treatment, as directed by their physician
* Pre-menopausal females and females < 2 years after the onset of menopause should have a negative pregnancy test at Screening. Pre-menopausal females must agree to use an acceptable method of birth control from the time of the negative pregnancy test up to 90 days after the last dose of the study drug
* Females of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for > 1 year
* Before study entry, written informed consent must be obtained from the patient prior to performing any study related procedures

Exclusion Criteria:

* Prior treatment with Vemurafenib or Dabrafenib
* Known hypersensitivity to Metformin or any of its components
* Received radiotherapy for non CNS disease within the 2 weeks prior to commencing study treatment or have not recovered from side effects of all radiation related toxicities to Grade < 1, except for alopecia
* Pregnant, breast feeding, or refusing double barrier contraception, oral contraceptives, or avoidance of pregnancy measures
* Have any other uncontrolled infection or medical condition that could interfere with the conduct of the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-17 (Actual)

PRIMARY OUTCOMES:
Observation of two CTCAE drug related grade 4 toxicities in six patients. | Duration of phase I portion, approxiately 6 months
  During phase I, six patients will be enrolled and monitored for toxicities. If drug related deaths occur or more than two drug related CTCAE grade 4 toxicities occur the trial will be suspended. Phase II will estimate the efficacy of the drugs, enrolling 20 patients during stage 1 with an upper limit of 39 for the 2nd stage.
Clinical Response Rate | 6 years
  Phase II will study the efficacy of the drugs enrolling 20 patients during stage I with an upper limit of 39 for the 2nd stage.

SECONDARY OUTCOMES:
To estimate the overall survival rates. | Approximately 3 years
  Patients will be contacted every 3 months following treatment administration for up to three years to obtain survival data.
To explore the effect of other covariates on overall survival | 3 years
  To identify demographic, disease and treatment related effects on overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Chesney, MD, PhD, Principal Investigator — James Graham Brown Cancer Center
Locations (2):
- United States (2):
  - James Graham Brown Cancer Center-Universityof Louisville, Louisville, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT02143050/Prot_SAP_000.pdf